CLINICAL TRIAL: NCT06034808
Title: Frequency of Sacroiliitis in Inflammatory Bowel Disease Patients Using MRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Magy Wageeh Abdelmalak, Director, Assiut University
Other Study IDs: Sacroliitis in IBD using MRI
Record Dates: First submitted 2023-09-02; First posted 2023-09-13 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Sacroiliitis
MeSH Terms: conditions — Sacroiliitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. to determine the overall frequency of Inflammatory sacroiliitis among patients with Inflammatory bowel disease using magnetic resonance imaging
2. identify the association of sacroliitis in IBD patients clinical and laboratory markers

DETAILED DESCRIPTION:
INFLAMMATORY BOWEL DISEASE (IBD) is a disorder in which an inappropriate response to an unknown antigen, combined with genetic and environmental factors, result in inflammation of the small bowel and colon . The two main forms of IBD are Crohn's disease (CD) and ulcerative colitis (UC) which are both associated with spondyloarthropathy (SpA), an inflammatory arthritis characterized by sacroiliitis and inflammatory back pain .

Articular manifestations of inflammatory bowel disease(IBD), comprising Crohn's disease (CD) and ulcerative colitis (UC), were first described in 1930 and have been considered as spondylarthropathies since 1978. They include peripheral arthritis and inflammatory axial involvement.

Extra-intestinal musculoskeletal manifestations associated with Inflammatory bowel disease, can be divided into axial and peripheral arthropathy, which can be a cause of significant morbidity that can adversely affect the quality of life in these patients. Peripheral arthropathy represent the most frequent (40%) extra-intestinal manifestation in IBD. These manifestations occur more frequently in patients with Crohn's disease.

Sacroiliitis (SI) is considered one of the common axial arthropathies with an estimated prevalence of around 10% of Crohn's patients.

It is crucial to differentiate inflammatory back pain due to axial SpA from other causes of chronic low back pain as they have different treatments and prognosis.

The diagnosis is based upon the presence of characteristic inflammatory type back pain with evidence of SI on imaging . Both clinical examination and plain radiographs have their own limitations of only detecting advanced disease.

Importantly, sacroiliitis, which is the hallmark of the spondyloarthropathies, may be clinically silent with an ambiguous or equivocal physical examination tests so imaginghas important role in its diagnosis Imaging findings in sacroiliitis are divided into acute and structural changes.The acute findings of sacroiliitis can be observed on magnetic resonance imaging (MRI) and include periarticular sacroiliac joint (SIJ) bone marrow edema(BME), soft tissue edema, and contrast enhancement. Structural changes including SIJ erosions, subchondral sclerosis and bony bridges appear relatively late in the disease .Indeed, findings compatible with acute inflammation may be seen on MRI years before late structural findings are evident.

MRI is a promising technology with a higher sensitivity and specificity for the diagnosis of SI. As MRI is being utilized more frequently in patients with Crohn's disease, more and more patients are found to have a positive MRI evidence of SI without clinical signs or symptoms so MRI is necessary for diagnosing and evaluating patients with early disease.

Incorporation of magnetic resonance imaging (MRI) to assess axial SpA allows early recognition of axial SpA in CD, especially when patients do not present with classic IBP symptoms.

The introduction of biological drugs from the tumor necrosis factor-alpha (TNF-a) receptor blocker group, has further emphasized the need for early diagnosis of sacroiliitis in patients with IBD, many of which, can be asymptomatic, nonradiographic, or both. These drugs, when administered early in the disease, are capable of changing the course, alleviating the symptoms and even producing withdrawal of early imaging findings, including BME and contrast enhancement.

ELIGIBILITY:
Inclusion Criteria:

* subjects between 18 and 65 years.
* subjects met clinical, pathological or radiological criteria of IBD.

Exclusion Criteria:

1. Patients who refuse enter the study
2. Patients who not diagnosed as IBD
3. other inflammatory arthritis (e.g. rheumatoid arthritis, systemic lupus erythematosus, psoriatic or reactive arthritis)
4. co-existent autoimmune diseases (e.g. celiac disease, Behcets disease)
5. malignancy less than 5 years in remission .
6. having a contraindication to MRI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients were selected from outpatient clinic of IBD of Elraghi hospital.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Primary (main) | through study completion, an average of 1 year
  Incidence of sacroliitis in inflammatory bowel disease patients using MRI
  with Inflammatory bowel disease using magnetic resonance imaging.

SECONDARY OUTCOMES:
Secondary | through study completion, an average of 1 year
  association of sacroliitis in IBD patients assessed by clinical and laboratory markers .
  * clinical examination including sacroiliac joint examination
  * Laboratory investigations

REFERENCES:
- [Background] Wills JS, Lobis IF, Denstman FJ. Crohn disease: state of the art. Radiology. 1997 Mar;202(3):597-610. doi: 10.1148/radiology.202.3.9051003. No abstract available.
- [Background] Leclerc-Jacob S, Lux G, Rat AC, Laurent V, Blum A, Chary-Valckenaere I, Peyrin-Biroulet L, Loeuille D. The prevalence of inflammatory sacroiliitis assessed on magnetic resonance imaging of inflammatory bowel disease: a retrospective study performed on 186 patients. Aliment Pharmacol Ther. 2014 May;39(9):957-62. doi: 10.1111/apt.12680. Epub 2014 Mar 4. PMID 24593050
- [Background] Veloso FT, Carvalho J, Magro F. Immune-related systemic manifestations of inflammatory bowel disease. A prospective study of 792 patients. J Clin Gastroenterol. 1996 Jul;23(1):29-34. doi: 10.1097/00004836-199607000-00009. PMID 8835896
- [Background] Sieper J, Rudwaleit M, Baraliakos X, Brandt J, Braun J, Burgos-Vargas R, Dougados M, Hermann KG, Landewe R, Maksymowych W, van der Heijde D. The Assessment of SpondyloArthritis international Society (ASAS) handbook: a guide to assess spondyloarthritis. Ann Rheum Dis. 2009 Jun;68 Suppl 2:ii1-44. doi: 10.1136/ard.2008.104018. PMID 19433414
- [Background] Oostveen J, Prevo R, den Boer J, van de Laar M. Early detection of sacroiliitis on magnetic resonance imaging and subsequent development of sacroiliitis on plain radiography. A prospective, longitudinal study. J Rheumatol. 1999 Sep;26(9):1953-8. PMID 10493676
- [Background] Sudol-Szopinska I, Urbanik A. Diagnostic imaging of sacroiliac joints and the spine in the course of spondyloarthropathies. Pol J Radiol. 2013 Apr;78(2):43-9. doi: 10.12659/PJR.889039. PMID 23807884
- [Background] Baraliakos X, van der Heijde D, Braun J, Landewe RB. OMERACT magnetic resonance imaging initiative on structural and inflammatory lesions in ankylosing spondylitis--report of a special interest group at OMERACT 10 on sacroiliac joint and spine lesions. J Rheumatol. 2011 Sep;38(9):2051-4. doi: 10.3899/jrheum.110423. PMID 21885516
- [Background] Bredella MA, Steinbach LS, Morgan S, Ward M, Davis JC. MRI of the sacroiliac joints in patients with moderate to severe ankylosing spondylitis. AJR Am J Roentgenol. 2006 Dec;187(6):1420-6. doi: 10.2214/AJR.05.1423. PMID 17114530
- [Background] Hermann KG, Bollow M. Magnetic resonance imaging of sacroiliitis in patients with spondyloarthritis: correlation with anatomy and histology. Rofo. 2014 Mar;186(3):230-7. doi: 10.1055/s-0033-1350411. Epub 2013 Sep 2. PMID 23999786
- [Background] Weber U, Lambert RG, Ostergaard M, Hodler J, Pedersen SJ, Maksymowych WP. The diagnostic utility of magnetic resonance imaging in spondylarthritis: an international multicenter evaluation of one hundred eighty-seven subjects. Arthritis Rheum. 2010 Oct;62(10):3048-58. doi: 10.1002/art.27571. PMID 20496416
- [Background] Baraliakos X, Listing J, Rudwaleit M, Haibel H, Brandt J, Sieper J, Braun J. Progression of radiographic damage in patients with ankylosing spondylitis: defining the central role of syndesmophytes. Ann Rheum Dis. 2007 Jul;66(7):910-5. doi: 10.1136/ard.2006.066415. Epub 2007 Feb 28. PMID 17329306
- [Background] van der Heijde D, Landewe R, Einstein S, Ory P, Vosse D, Ni L, Lin SL, Tsuji W, Davis JC Jr. Radiographic progression of ankylosing spondylitis after up to two years of treatment with etanercept. Arthritis Rheum. 2008 May;58(5):1324-31. doi: 10.1002/art.23471. PMID 18438853